CLINICAL TRIAL: NCT05614336
Title: Corona-Virus-Disease 2019 (Covid-19) Antibody Responses in Cystic Fibrosis
Brief Title: COVID-19 Antibody Responses in Cystic Fibrosis
Acronym: CAR-CF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_0478
Record Dates: First submitted 2022-11-10; First posted 2022-11-14 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Cystic Fibrosis
MeSH Terms: conditions — COVID-19; Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cystic Fibrosis patients (Other): Patients with cystic fibrosis, regardless of age, genetic profile, transplant status and disease severity will be eligible to participate in the study.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood serum samples will be collected for analysis of COVID-19 antibody levels. For participants who consent to the optional study, a second blood sample will also be drawn into EDTA tubes (plasma)

SUMMARY:
Coronavirus disease 2019 (COVID-19) which is caused by the virus SARS-CoV-2 has resulted in an ongoing global pandemic. It is unclear whether the relatively low number of reported cases of COVID-19 in people with CF (pwCF) is due to enhanced infection prevention practices or whether pwCF have protective genetic/immune factors. This study aims to prospectively assess the proportion of pwCF, including both adults and children with CF who have evidence of SARS-CoV-2 antibodies over a two-year period. This study will also examine whether pwCF who have antibodies for SARS-CoV-2 have a different clinical presentation and what impact this has on their CF disease. The proposed study will recruit pwCF from paediatric and adult CF centres in Europe. Serological testing to detect antibodies will be performed on blood samples taken at month 0, 6, 12, 18 and 24 with additional time-points if bloodwork is available via normal clinical care. Clinical data on, lung function, CF-related medical history, pulmonary exacerbations, antibiotic use, and microbiology and vaccination receipt, will be collected during routine clinical assessments. Associations will be examined between socio-demographic and clinical variables and serologic testing. The effects of SARS-CoV-2 infection on clinical outcomes and analyse end-points will be examined to explore any age-related or gender-based differences, as well as subgroup analysis of outcomes in lung-transplant recipients and pwCF receiving CFTR modulator therapies. As pwCF receive COVID-19 vaccination a comparison of the development and progression of anti-SARS-CoV-2 antibodies in pwCF following natural infection and vaccination SARS-CoV-2 over time will be performed

ELIGIBILITY:
Inclusion Criteria:

* Person with cystic fibrosis of any age, genotype, transplant status and disease severity.
* Express consent obtained after informing the patient and/or his legal representatives or parents In France, written and informed consent will be requested.
* For France, affiliation to a social security scheme or similar

Exclusion Criteria:

* Refusal to give informed consent
* Contraindication to venepuncture
* For France

  * Person under guardianship / curatorship
  * Person under legal protection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
SARS-COV-2 seroprevalence | 2 years
  Proportion of pwCF with at least 1 seropositive result over the study period and the difference in this proportion by age, geographical area and over time.

SECONDARY OUTCOMES:
Association of SARS-CoV-2 seropositivity, clinical symptoms and clinical outcomes in pwCF | 2 years
  Incidence of symptomatic COVID-19 over the study period and severity; proportion of seropositive pwCF with subsequent CF exacerbation compared to pwCF who are seronegative; death rate in pwCF with at least one seropositive result compared to pwCF who are seronegative.
Longitudinal comparison of the detection including level and duration of anti-SARS-CoV-2 antibodies in pwCF following natural infection and SARS-CoV-2 vaccination | 2 years
  Longitudinal comparison of the detection including level and duration of anti-SARS-CoV-2 antibodies in pwCF following natural infection and SARS-CoV-2 vaccination
Serum proteomic and genomic responses of pwCF who are SARS-CoV-2 seropositive an seronegative | 10 years maximum
  Serum proteomic and genomic responses of pwCF who are SARS-CoV-2 seropositive an seronegative

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - C.R.C.M. Pédiatrique (Centre de Ressources et de Compétences en Mucoviscidose) Hôpital des Enfants-Pellegrin - CHU de Bordeaux, Bordeaux
  - Pneumologie, allergologie et Mucoviscidose - CRCM Lyon pédiatrie Hôpital Femme Mère Enfant /Groupement Est, Bron
  - Centre de Ressources et de Competences de la Mucoviscidose (Enfants) CHU Grenoble Alpes - Hôpital Couple Enfant, Grenoble
  - Service des maladies respiratoires Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier
  - Service de pédiatrie générale et spécialisée American Memorial Hospital - CHU de Reims, Reims
  - Fondation Ildys, Roscoff
  - Maladies respiratoires, allergologie - CRCM Mixte de Rouen Hôpital Charles Nicole - CHU de Rouen, Rouen
  - Service de pneumo-allergologie pédiatrique CRCM pédiatrique CHU de Toulouse - Hôpital des Enfants, Toulouse
  - Service Pneumologie-Allergologie CRCM adulte Hôpital Larrey - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No